CLINICAL TRIAL: NCT02469519
Title: A Randomized Double-blinded Trial Comparing the Impact of One Versus Two Courses of Antenatal Steroids on Neonatal Outcome in the Patient With Prelabor Premature Rupture of the Membranes
Brief Title: Impact of a Booster Course of Antenatal Steroids on Neonatal Outcome in Patients With Premature Rupture of the Membranes
Acronym: ACSinPROM
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pediatrix (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OBX0034
Record Dates: First submitted 2015-06-05; First posted 2015-06-11 (Estimated); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Premature Birth
MeSH Terms: conditions — Premature Birth | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Betamethasone - ACTIVE (Experimental): Booster Course of Antenatal Steroids consists of Betamethasone [12 mg intramuscular injection, 24 hours apart X 2 doses] or if unavailable may give Dexamethasone [6 mg intramuscularly 12 hours apart x 4 doses]
  Interventions: Drug: Betamethasone - ACTIVE
- normal saline - PLACEBO (Placebo Comparator): Normal saline of equivalent volume given intramuscularly at the equivalent dosing regimes listed in experimental arm.
  Interventions: Other: Normal Saline - PLACEBO

INTERVENTIONS:
Drug: Betamethasone - ACTIVE — antenatal corticosteroid (ACS) is to be given by injection 24 hours apart for two doses.
  Other Names: antenatal corticosteroid; dexamethasone
  Arms: Betamethasone - ACTIVE
Other: Normal Saline - PLACEBO — normal saline of the same quantity as with the experimental drug is to be given by injection 24 hours apart for two doses
  Other Names: NS
  Arms: normal saline - PLACEBO

SUMMARY:
This trial hopes to prospectively evaluate the impact of one versus two courses of antenatal steroids on the incidence of major neonatal morbidity in pregnant women with pre-labor premature rupture of the membranes.

DETAILED DESCRIPTION:
This is a multicenter randomized double blinded trial that hopes to prospectively evaluate the impact of one versus two courses of antenatal steroids on the incidence of major neonatal morbidity including respiratory distress syndrome in pregnant women with a singleton gestation between 24w0d - 32w6d gestation who have documented premature rupture of the membranes.

ELIGIBILITY:
Inclusion Criteria:

* Participants age 18 years or older
* 24w0d to 32w6d weeks gestation
* Singleton pregnancy
* Received first course of ACS at or prior to 31w6d gestation
* Began first course of ACS at least 7 days ( =/> 168 hours) prior to randomization
* Expectant management planned
* Premature Ruptured membranes (PROM) before onset of labor

Exclusion Criteria:

* Known major fetal anomalies
* Multiple gestation
* Not a candidate for expectant management
* Clinical chorioamnionitis (two or more of the following: temperature > 38.0 degrees centigrade; uterine tenderness; foul smelling vaginal discharge or amniotic fluid; maternal tachycardia >100 bpm; fetal tachycardia >160 bpm; maternal White Blood Cell (WBC) count >20 X 109/L; C-Reactive Protein (CRP) > 5.9
* Already receiving corticosteroids for another condition
* Any contraindications to the maternal use of corticosteroids

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2016-03-03 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Composite Neonatal Morbidity | from birth through the first 28 days of life
  Composite Neonatal Morbidity includes any one or more of the following: respiratory distress syndrome, bronchopulmonary dysplasia, severe intraventricular hemorrhage, periventricular leukomalacia, proven sepsis, necrotizing enterocolitis, or neonatal death.

SECONDARY OUTCOMES:
Gestational age of baby | measured within the first 24 hours following birth.
  gestational age of the baby on the day of it's birth
Baby's birth weight | measured within the first 24 hours following birth
  weight of the baby taken with in the first hours following birth
Intrauterine growth restriction (IUGR) | anytime during the pregnancy prior to birth (~ 9 months of pregnancy)
  a measurement done by ultrasound taken at any time during the pregnancy prior to birth
Baby's Head Circumference | measured within the first 24 hours following birth
  a measurement of the baby's head taken within the first hours following birth
Newborn Mechanical Ventilatory days | measured from birth to 28 days following birth
  measurement of the total number of days the baby requires mechanical ventilatory support
Newborn Oxygen support days | measured from birth to 28 days following birth
  measurement of the total number of days the baby requires oxygen support (example: nasal cannula, CPAP)
Newborn Surfactant therapy | measured within the first 24 hours following birth
  measurement of the need for newborn surfactant therapy within the first 28 day following birth
Newborn Hospital Days | measured within the first 24 hours following birth
  the number of days that newborn remains in the hospital following its birth.
Pneumothorax | measured within the first 24 hours following birth
  diagnosis of a collapsed lung supported by clinical or radiologic evidence.
Maternal Infectious Morbidity | measured within the first 24 hours following birth
  diagnosis of maternal infection for example; chorioamnionitis, endometritis or postoperative wound infection.
time from first dose of study drug to birth | measured in days/hours from the time of administration of first study drug until birth.
  the number of hours/days from the time of the first dose of study drug until birth

CONTACTS AND LOCATIONS:
Overall Officials: Richard Porreco, MD, Principal Investigator — Pediatrix
Locations (9):
- United States (9):
  - University of South Alabama Medical Center, Mobile, Alabama
  - Phoenix Perinatal Associates, Phoenix, Arizona
  - Long Beach Memorial Medical Center, Long Beach, California
  - Good Samaritan Hospital, San Jose, California
  - Presbyterian/St Luke's Hospital, Denver, Colorado
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Lousiana State University Health Science, Shreveport, Louisiana
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Swedish Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Porreco R, Garite TJ, Combs CA, Maurel K, Huls CK, Baker S, Fortner KB, Longo SA, Nageotte M, Lewis D, Tran L; Obstetrix Collaborative Research Network. Booster course of antenatal corticosteroids after preterm prelabor rupture of membranes: a double-blind randomized trial. Am J Obstet Gynecol MFM. 2023 May;5(5):100896. doi: 10.1016/j.ajogmf.2023.100896. Epub 2023 Feb 14. PMID 36796641